CLINICAL TRIAL: NCT00907257
Title: A Clinical Assessment of the Use of RETIN-A MICRO (Tretinoin Gel) Microsphere, 0.04% in a Pump Dispenser and a 5% Benzoyl Peroxide Wash Used in the Morning Compared to the Use of RETIN-A MICRO 0.04% Pump Nightly and a 5% Benzoyl Peroxide Wash in the Morning For the Treatment of Facial Acne Vulgaris
Brief Title: A Study of Different Use Regimens Using Two Acne Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CA-P-6270
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: acne; irritation; objective sensory methods
MeSH Terms: conditions — Acne Vulgaris | interventions — Triclosan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Same time of day (Experimental): 5% benzoyl peroxide wash and 0.04% tretinoin gel used at same time of day
  Interventions: Drug: benzoyl peroxide wash; Drug: Tretinoin gel
- Different times of day (Active Comparator): 5% benzoyl peroxide wash used in the morning and 0.04% tretinoin gel used in the evening
  Interventions: Drug: benzoyl peroxide wash; Drug: Tretinoin gel

INTERVENTIONS:
Drug: benzoyl peroxide wash — 5% benzoyl peroxide wash
  Other Names: OXY Wash
Drug: Tretinoin gel — 0.04% tretinoin gel
  Other Names: Retin-A Micro Pump

SUMMARY:
A study to determine if using 2 acne products in the morning is as safe and efficacious as using one product in the morning and one product in the evening.

DETAILED DESCRIPTION:
Approximately 240 subjects will be enrolled in this randomized, multi-center study. Following satisfaction of entry criteria and screening procedures, all subjects will receive RETIN-A MICRO PUMP 0.04% and a 5% Benzoyl Peroxide wash (OTC) for the entire 12-week treatment period. Subjects will be randomized to either both morning treatments (test) or to the morning/evening treatment (active control). Subjects will be assessed at baseline, at week 3, week 6 and again at the end of therapy, week 12 for number and type of individual lesions and safety. At selected sites, photographs will be taken at the same time points. At Week 12 subjects will be assessed for Investigator's Global Assessment of Acne Severity. The investigator will conduct all of the lesion counts, global assessments and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant or non-nursing females, 12 years or older, with facial acne vulgaris;
* Minimum of 20 but no more than 50 inflammatory lesions (papules and pustules);
* Minimum of 30 but no more than 100 facial non-inflammatory lesions (open and closed comedones);
* Must have at least a rating of grade 3 on the Investigator Global severity scale at baseline

Exclusion Criteria:

* Known sensitivity to any of the ingredients in the study medication;
* Any nodulocystic acne lesions;
* Use of acne devices or systemic therapy with antibiotics within two months prior to start and throughout the duration of the study;
* Use of systemic therapy with retinoids within four months prior to study start and throughout the duration of the study;
* Topical use of retinoids within two weeks prior to study start and throughout the duration of the study;
* Topical use of antibiotics, steroids and/or other non-retinoid topical acne products within two weeks prior to study start and throughout the duration of the study;
* If subject is taking birth control pills, she must be stabilized for at least three months prior to study start;
* History of evidence of other skin conditions or diseases that may require concurrent therapy or may interfere with the evaluation of the study medication;
* Any significant medical conditions that could confound the interpretation of the study;
* Excessive facial hair that may interfere with evaluations;
* No use of tanning booths, sun lamps, etc.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rossi, MD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (12):
- United States (12):
  - Skin Care Research, Inc., Boca Raton, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Gwinnett Clinical Research, Snellville, Georgia
  - Derm Research, PLLC, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - DermResearch Center of New York, Stony Brook, New York
  - Dermatology Research Associates, Cincinnatti, Ohio
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - DermResearch, Inc., Austin, Texas
  - Education & Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- [Result] Pariser D, Bucko A, Fried R, Jarratt MT, Kempers S, Kircik L, Lucky AW, Rafal E, Rendon M, Weiss J, Wilson DC, Rossi AB, Ramaswamy R, Nighland M. Tretinoin gel microsphere pump 0.04% plus 5% benzoyl peroxide wash for treatment of acne vulgaris: morning/morning regimen is as effective and safe as morning/evening regimen. J Drugs Dermatol. 2010 Jul;9(7):805-13. PMID 20677537
- See also: FDA's Drug Finder — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Same Time of Day | Different Times of Day
Started | 123 | 124
Completed | 110 | 112
Not Completed | 13 | 12
Not completed — Adverse Event | 0 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Per IRB-Subject became vulnerable | 1 | 0
Not completed — Moved | 1 | 0
Not completed — Personal Reasons | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Same Time of Day | Different Times of Day | Total
Number analyzed (Participants) | 123 | 124 | 247
Age Continuous [Mean (Standard Deviation); unit: years] | 18.5 (6.86) | 18.6 (6.94) | 18.5 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 66 | 126
  Male | 63 | 58 | 121
Region of Enrollment [Number; unit: participants]
  United States | 123 | 124 | 247
Fitzpatrick Score [Number; unit: Participants] — Skin type is categorized according to the Fitzpatrick skin type scale, which ranges from very fair (skin type I) to very dark (skin type VI).
  Participants
    I | 8 | 5 | 13
    II | 31 | 29 | 60
    III | 44 | 52 | 96
    IV | 24 | 22 | 46
    V | 8 | 12 | 20
    VI | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Facial Acne Lesion Count
Description: Total Facial Acne Lesion Count is the sum of non-inflammatory and inflammatory lesions, plus nodules/cysts. Change from Baseline is calculated as the value after Baseline minus the baseline value, and negative values indicate improvement.
Time Frame: Baseline to Week 12
Population: Per Protocol Population, which includes all Intention to Treat (ITT) subjects who completed the 12 weeks of treatment and evaluations with no major protocol deviations.
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Same Time of Day | Different Times of Day
Number analyzed (Participants) | 109 | 112
Lesions | 39.74 (1.64) | 40.02 (1.62)

2. Secondary Outcome: Change From Baseline in Inflammatory and Non-Inflammatory Lesion Counts and Their Totals
Description: Between group comparison with Last Count Carried Forward (LOCF) of Inflammatory Facial Acne Lesion Count (the sum of papules and pustules), Non-Inflammatory Facial Acne Lesion Count (the sum of open and closed comedones), and their Total (the sum of Non-inflammatory and Inflammatory lesions).
Time Frame: Baseline to Week 12
Population: Data set includes all Intent to Treat (ITT)subjects. Imputation technique was Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Same Time of Day | Different Times of Day
Number analyzed (Participants) | 123 | 124
Lesions
  Inflammatory Lesions | 14.6 (0.85) | 14.2 (0.84)
  Non-Inflammatory Lesions | 23.2 (1.17) | 23.7 (1.16)
  Total Lesions | 37.4 (1.70) | 38.1 (1.68)

3. Secondary Outcome: Measurement of Success
Description: Number of subjects achieving success according to dichotomized Investigator Global Assessment (IGA) using criteria of grades 0 or 1, or improvement of 2 grades from baseline score. Possible grades from 0-6 are described as follows:
  0 = Clear, 1=Almost Clear, 2=Mild, 3=Mild to Moderate, 4=Moderate, 5=Moderately Severe, 6=Severe.
Time Frame: Baseline to Week 12
Population: Intention to Treat (ITT)population and imputation technique of Last Observations Carried Forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Same Time of Day | Different Times of Day
Number analyzed (Participants) | 123 | 124
Participants
  Clear / Almost Clear | 26 | 25
  Improved Two Categories | 51 | 54

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Same Time of Day | Different Times of Day
Serious Adverse Events (participants affected / at risk) | 3/123 | 0/124
Other Adverse Events (participants affected / at risk) | 0/123 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Same Time of Day (N=123) | Different Times of Day (N=124)
Cardiac Arrhythmia (Cardiac disorders) | 1 | 0
Viral Myocarditis (Cardiac disorders) | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less